CLINICAL TRIAL: NCT04327999
Title: Effect of Artificial Tears on Radioiodine Levels in the Nasolacrimal Duct System of Patients Following Radioiodine Therapy for Thyroid Carcinoma
Brief Title: Effect of Artificial Tears on Radioiodine Levels in the Nasolacrimal Duct System
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Funding ended
Sponsor: Vanderbilt-Ingram Cancer Center (Other)
Responsible Party: Principal Investigator, Rachel Sobel, Principal Investigator, Vanderbilt-Ingram Cancer Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: VICC HN 2018
Record Dates: First submitted 2020-03-04; First posted 2020-03-31 (Actual); Results first posted 2024-01-18 (Actual); Last update posted 2024-01-18 (Actual); Status verified 2024-01

CONDITIONS: Thyroid Carcinoma; Radioactive Iodine Level
MeSH Terms: conditions — Thyroid Neoplasms | interventions — Lubricant Eye Drops

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Preservative free artificial tears (Experimental): Day 1, patients will self-administer artificial tears every 15 minutes for 2 hours followed by every 30 minutes for at least 4 hours or until bedtime at night. On Day 2, patients will self-administer artificial tears every 1 hour for 12 hours. On Day 3, patients will self-administer artificial tears four times that day. On Day 4, patients will self-administer tears twice that day. Patients will be instructed to wear their contact lenses throughout their waking hours.
  Interventions: Drug: Artificial Tears

INTERVENTIONS:
Drug: Artificial Tears — Self-Administered - utilizing eye drop preservative free vials

SUMMARY:
The purpose of this study is to explore whether administration of preservative free artificial tears will decrease the level of detectable radioiodine in the tears and nasolacrimal duct system of patients undergoing radioiodine therapy for thyroid carcinoma and thus decrease the risk of developing radioactive iodine associated nasolacrimal duct obstruction.

DETAILED DESCRIPTION:
Primary Objective:

- To assess whether use of preservative free artificial tears following radioactive iodine administration will lower the level of radioactive iodine in the tears of patients treated with radioactive iodine for thyroid carcinoma.

Secondary Objective:

- To evaluate whether artificial tears would be an effective preventative intervention to decrease the risk of developing nasolacrimal duct stenosis, which has been associated with radioactive iodine administration.

ELIGIBILITY:
Inclusion Criteria:

* Radio-iodine therapy for thyroid cancer
* Radioiodine therapy ≥100mCi
* Patient wears soft contacts on both eyes

Exclusion Criteria:

* Use of eye drops, other than artificial tears
* History of periocular trauma with tear duct involvement/lacrimal gland trauma
* History of lacrimal drainage disease: canaliculitis, dacryocystitis
* Prior radiotherapy
* Current or prior use of chemotherapy drugs (i.e. 5-fluorouracil, docetaxel)
* Medical conditions that predispose to NLD stenosis

  * Sarcoid
  * Granulomatosis with polyangiitis
  * Chronic lymphocytic leukemia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2020-10-05 (Actual); Primary Completion 2023-09-25 (Actual); Study Completion 2023-09-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rachel Sobel, MD, Principal Investigator — Vanderbilt Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

REFERENCES:
- [Derived] Lee IT, Grice JV, Ji X, Chen Q, Bischoff LA, Jessop AC, Barahimi B, Codere F, Mawn LA, Sobel RK. A Pilot Nonrandomized Controlled Trial Examining the Use of Artificial Tears on the Radioactivity of Tears After Radioactive Iodine Treatment for Thyroid Cancer. Thyroid. 2024 Jan;34(1):82-87. doi: 10.1089/thy.2023.0338. Epub 2023 Dec 11. PMID 37917111

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Preservative Free Artificial Tears
Started | 9
Completed (1 patient was excluded for deviation from protocol) | 8
Not Completed | 1
Not completed — Protocol Violation | 1

BASELINE CHARACTERISTICS:
Arm/Group | Preservative Free Artificial Tears
Number analyzed (Participants) | 9
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 8
  >=65 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 5
  Unknown or Not Reported | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 7
  More than one race | 0
  Unknown or Not Reported | 2
Region of Enrollment [Number; unit: participants]
  United States | 9

OUTCOME MEASURES:

1. Primary Outcome: Change in Level of Radioactive Iodine in Tears
Description: The radioactive iodine activity level in the tears will be measured, as collected via contact lenses. Each patient will have a control eye and an experimental eye that received artificial tears. The control eye has no intervention. The radioactive iodine activity level will be measured over four days, with Day 1 occurring on the Day of systemic radioactive iodine therapy. On each of the four days, the level of radioactive iodine will be compared between the control and experimental eyes to see if there is a statistical difference between the control and experimental eyes.
Time Frame: Over a 4 day period
Measure: Geometric Mean (95% Confidence Interval); unit: Becquerel
Arm/Group | Preservative Free Artificial Tears
Number analyzed (Participants) | 8
Becquerel | 2975.7 [1579 to 5609]

ADVERSE EVENTS:
Time Frame: Approximately 32 months and 15 days.
Arm/Group | Preservative Free Artificial Tears
All-Cause Mortality (participants affected / at risk) | 0/9
Serious Adverse Events (participants affected / at risk) | 0/9
Other Adverse Events (participants affected / at risk) | 1/9
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Preservative Free Artificial Tears (N=9)
Early vasovagal response (Nervous system disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-04-17): https://cdn.clinicaltrials.gov/large-docs/99/NCT04327999/Prot_SAP_002.pdf
  • Informed Consent Form (2022-03-08): https://cdn.clinicaltrials.gov/large-docs/99/NCT04327999/ICF_001.pdf